CLINICAL TRIAL: NCT02403973
Title: Randomized Clinical Trial Comparing Perioperative Care for Breast Cancer Patients at a Patient Hotel Versus a General Surgical Ward
Brief Title: Trial Comparing Perioperative Care for Breast Cancer Patients at a Patient Hotel vs a General Surgical Ward
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danderyd Hospital (Other)
Collaborators: Indikator - Institutet för kvalitetsindikatorer (Unknown)
Responsible Party: Principal Investigator, Madleen Huzell, M.D., Danderyd Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2010/38-31/4
Record Dates: First submitted 2015-03-17; First posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer
Keywords: Patient hotel; Patient Satisfaction; Perioperative care; IN2005E
MeSH Terms: conditions — Breast Neoplasms; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient hotel group (Other)
  Interventions: Other: IN2005E
- Ward group (Other)
  Interventions: Other: IN2005E

INTERVENTIONS:
Other: IN2005E — IN2005E is a validated questionnaire that measures patient satisfaction

SUMMARY:
To explore the possible benefit of a patient hotel, a study was undertaken to test the hypothesis that perioperative care at a patient hotel would be valued better than care in a general ward. The study focuses solely on the patients' perspective and satisfaction of the care provided.

DETAILED DESCRIPTION:
The study was designed as a prospective randomised controlled trial, carried out at a single centre (Danderyds University Hospital). The protocol was approved by the Ethical committee for human studies.

With a primary outcome that perioperative care at the hotel would be valued 15-20% higher than care in a general ward, a power analysis, two-sided with α = 0.05, indicated that a sample size of 150 was needed to attain a power of 80%.

The patients were randomised to receive pre- and postoperative care either in a general surgical ward or at a patient hotel by using a sealed envelope method.

To evaluate the patients' experiences of the care provided at the ward and the hotel, respectively, the Swedish validated version of the adult inpatient survey of 2005 (IN2005-E) was used.

Adjacent to the discharge from the ward or hotel, the patient was provided with the IN2005-E questionnaire, which was filled out before the patient left the facility. The filled out form was sealed in an envelope by the patient herself and thereafter sent to a separate institute (Indikator) for further analysis. Indikator is responsible for the majority of the statistical analysis of patient surveys in Sweden.

Patient characteristics were compared using a confidence interval of 95%. The SF-36 was analyzed with a two-sample t-test. The IN2005E was analyzed by a cross-tabulation of the data using the χ² test in SPSS 17.0. The significance level was set to < 0.05.

ELIGIBILITY:
Inclusion Criteria:

Women with a breast tumour, who were to undergo surgical treatment in order to remove a known cancer or to exclude cancerous changes in a diagnosed tumour

Exclusion Criteria:

* Insulin dependent diabetes
* Severe impairment of mobility
* A known coagulopathy
* Cancer surgery with a coherent primary reconstruction
* Severe cardiac illness
* An inability to understand Swedish
* Mental incapacity.

Max Age: 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2010-04; Primary Completion 2012-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction regarding provided care associated with surgery for breast cancer | in average 1 day
  The IN2005-E is a quantitative questionnaire, based upon the Picker Adult Inpatient Questionnaire and is commonly used to examine specific aspects of patient satisfaction. The IN2005-E is comprised by questions that focus on whether a specific event occurred or not, rather than letting the patients rate their care in terms of how satisfied they are. By this design the influence of outside factors is reduced. The conceptual basis and design of the original questionnaire has been described in detail elsewhere (Cleary PD, Edgman-Levitan S, Roberts M, Moloney TW, McMullen W, Walker JD, Delbanco TL. "Patients evaluate their hospital care: a national survey". Health Affairs 1991; 10; 254-267. Cleary PD, Edgman-Levitan S, Walker JD, Gerteis M, Delbanco TL. "Using patient reports to improve the medical care: a preliminary report from 10 hospitals". Quality Management in Health Care 1993; 2: 31-8. http://nhssurveys.org/surveys/712)